CLINICAL TRIAL: NCT02954861
Title: A Study to Identify the Incidence of Post Traumatic Stress Symptoms in Patients With Delirium Following Cardiac Surgery
Status: Completed | Type: Observational
Sponsor: University of Edinburgh (Other)
Collaborators: NHS Lothian (Other Government)
Responsible Party: Sponsor
Other Study IDs: 172976
Record Dates: First submitted 2016-09-08; First posted 2016-11-04 (Estimated); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Cardiac Disease; Delirium; Stress Disorders, Post-Traumatic
MeSH Terms: conditions — Heart Diseases; Delirium; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Cardiac surgery: Patients who develop delirium following cardiac surgery
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
'Post perfusion syndrome' was a term historically associated to cardiac surgery in view of the transient neuro-cognitive deficits attributed to cardio pulmonary bypass pump. During their recovery period, a significant number of patients experience delirium, a clinical syndrome of acute onset and fluctuant course.Though these deficits are often known to be transient without any permanent physical or neurological impairment, the experience can still psycho-socially affect these patients for a longer length of time even after discharge. The presence of delirium puts excessive, undesired strain on the patient, their families, health care providers and hospital resources.

PTSS is an anxiety disorder caused by very stressful, frightening or distressing events. It is known to either develop immediately after the disturbing event or weeks and months later. The actual symptoms can be varied but are categorized in three sections: i.e.: re-experiencing, avoidance and emotional numbing and hyperarousal (feeling 'on edge').

A problem that has such an impact on any patient is worth investigating and understood better. Being in such a unique professional position, as a Clinical nurse practitioner, the investigator is ideally placed to conduct this study. In this study, the researcher will be focusing on the pre-operative risk factors in developing delirium, actual incidence of delirium and follow the patients post operatively to evaluate the after effects of delirium in the form of PTSS.

DETAILED DESCRIPTION:
Delirium is acute onset of fluctuant cognitive state. Post operative delirium is a historically known complication after cardiac surgery. In 2013, almost 900 heart operations were performed in a South East, Scottish Cardio Thoracic unit. and audit data shows that 45% of these patients developed post operative delirium.

Multiple pre, post & intra operative factors have been attributed to the development of delirium. Whatever the precipitating factors, delirium not only causes psychological distress to the patient but also their loved ones. In some cases this psychological upset continues to affect the patient even after discharge from the hospital referred to as post traumatic stress symptoms (PTSS). This study therefore aims to look at the extent and experience of post operative delirium in cardiac surgery patients.

The study plans to recruit patients at a pre admission clinic where patient's baseline clinical data will be collected. They will also be provided with questionnaires to complete before the end of the clinic. This is to evaluate the participant's pre operative mood, cognitive status and social orientation. During their hospital stay following surgery the participants will be assessed routinely for delirium. If they are known to have suffered from delirium, they will be enrolled to phase 2 of the study.

The consented patients will be seen at 6 week follow up clinic where they will be provided with a questionnaire to identify PTSS and also participate in a semi structured interview. Three months later the same will be repeated on telephone.

Data analysis will help understand and explore this unfortunate patient experience.

ELIGIBILITY:
The target population will be all consecutive patients being operated during the data collection period.

Inclusion criteria:

* Male or female participants age 18 and over.
* Adults with capacity to informed consent
* Elective and urgent conventional cardiac surgery.

Exclusion Criteria:

* Patients from the highlands and islands who may not wish to return to the 6 weeks follow up clinic
* Re-do Cardiac surgery
* Emergency Cardiac surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Following discussion with statisticians and viewing the sample sizes of previous related studies, it was suggested that minimum 200 patients will be required for phase I. This was based on the availability of data in a similar aspects of the study. But incidentally there has been no known study looking specifically at delirium and post traumatic stress symptoms in cardiac surgery patients. So the researcher aims to enrol at least 400 patients but may not be able to achieve this number by the end of data collection phase.
  Phase II will only have patients who develop delirium and convenient sampling will be applied for the interview section.
Sampling Method: Probability Sample
Enrollment: 406 (Actual)
Dates: Start 2016-04-07 (Actual); Primary Completion 2018-03-30 (Actual); Study Completion 2018-05-10 (Actual)

PRIMARY OUTCOMES:
What factors during the peri-operative period in patients with delirium are associated with higher incidence of post traumatic stress symptoms? | 6 weeks and 3 months following delirium post cardiac surgery

SECONDARY OUTCOMES:
What are the peri-operative factors that are associated with change in PTSS score from 6 weeks to 3 months. | 6-12 weeks
What are the pre operative features that predict post operative delirium | 5 days
  The pre operative data collected will form an entry baseline for the study. But this will also aid in identifying common factors that are noted in patients who develop post operative delirium.

IPD SHARING:
Plan to Share IPD: No